CLINICAL TRIAL: NCT00922155
Title: Clinical Effectiveness of a Balloon Covered Sheath as a Guide Sheath in Endobronchial Ultrasound Guided Diagnosis of Peripheral Lung Lesions
Brief Title: Diagnosis of Lung Lesions by Endobronchial Ultrasound With an Alternative Guide Sheath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Yung-Lun Ni, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 96-0011B
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2007-03

CONDITIONS: Pulmonary Neoplasms; Solitary Pulmonary Nodules
Keywords: endobronchial ultrasound; guide sheath; peripheral pulmonary lesions
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBUS (No Intervention): After the PPLs been localized by endobronchial ultrasound(EBUS), patients in the EBUS group received transbronchial biopsy and bronchial washing at the bronchus located by EBUS.
- EBUS-GS (Active Comparator): After PPLs been localized by EBUS, the EBUS and guide sheath were then inserted to localize the lesion again. Transbronchial biopsy and brushing were done through the guide sheath after the probe been removed.
  Interventions: Device: guide sheath

INTERVENTIONS:
Device: guide sheath — The guide sheath (GS) was originally the balloon covered sheath (MAJ-643R, external diameter 2.6mm) of the EBUS probe. The two ends of the balloon covered sheath were cut and trimmed. The EBUS probe was covered with guide sheath and then inserted through the working channel to the targeted bronchus.
  Arms: EBUS-GS

SUMMARY:
The purpose of this study is to examine the usefulness of a balloon covered sheath as a guide sheath in endobronchial ultrasound guided transbronchial biopsy and bronchial brushing cytology for diagnosis of peripheral lung lesions

DETAILED DESCRIPTION:
Flexible bronchoscopy has been applied in the diagnosis of peripheral pulmonary lesions (PPLs) for decades. Without accurate localization, the diagnostic yield for peripheral lung cancers by these procedures is limited and variable. Localization of peripheral lung cancers can be aided by the use of computed tomography or fluoroscopy during fiberoptic bronchoscopy. However, radiation exposure to staffs and patients is always a concern in these procedures.

The clinical application of endobronchial ultrasound (EBUS) included determination of the depth of tumor invasion in tracheobronchial wall, evaluation of tracheobronchial structure before therapeutic bronchoscopy, localization of site of biopsy, EBUS-guided transbronchial needle aspiration, and analysis of peripheral tumor. Under EBUS guidance, the diagnostic yield of transbronchial lung biopsy in patients with peripheral lung cancer by bronchoscopic examination was significantly improved without an increase in the complication rate. More recently, with the aid of a guide sheath (EBUS-GS), EBUS has been shown to increase the diagnostic yield of PPLs, even in patients with fluoroscopy-invisible lung nodules, and avert the need for surgical procedures.

Most recently used GS for EBUS are specified for the EBUS probe with an external diameter of 1.9 mm. Such a thin caliber GS is designed to reach the PPLs, sometimes with an aid of curette, to provide an exact site for repeated obtainment of adequate specimens. We wonder whether a larger caliber sheath transformed from a balloon covered with an external diameter of 2.6 mm without reaching the PPLs, can offer similar effectiveness in diagnosis of the PPLs. The results may provide an alternative way for EBUS-GS especially in those countries where the commonly used GS of EBUS is not available.

ELIGIBILITY:
Inclusion Criteria:

* patients with peripheral pulmonary lesions who are going to receive bronchoscopy

Exclusion Criteria:

* endobronchial abnormalities
* associated lung parenchyma changes, ex. lung collapse or atelectasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
the diagnostic efficiency of flexible bronchoscopy(FB) in peripheral lung lesions(PPLs) | 1 year

SECONDARY OUTCOMES:
complications, including bleeding, pneumothorax, respiratory failure, | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department or Chest Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan